CLINICAL TRIAL: NCT04493463
Title: Effects of Methylprednisolone Plus Ropivacaine Infiltration Before Wound Closure on Laminoplasty or Laminectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY 2019-112-02-2
Record Dates: First submitted 2020-07-26; First posted 2020-07-30 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain; Neurosurgery
Keywords: Postoperative Pain; Methylprednisolone; Ropivacaine; Local Infiltration; Laminoplasty; Laminectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Methylprednisolone; Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- methylprednisolone + ropivacaine + saline (Experimental): The local infiltration solution in the methylprednisolone plus ropivacaine with saline group (treatment group) will consist of 1 ml of 40 mg methylprednisolone plus 15ml of 1% ropivacaine and 14 ml saline.
  Interventions: Drug: Methylprednisolone 40 mg + Ropivacaine + Saline
- ropivacaine + saline (Active Comparator): The local infiltration solution in the ropivacaine plus saline group (control group) will consist of 15 ml of 1% ropivacaine and 15ml saline.
  Interventions: Drug: Ropivacaine + Saline

INTERVENTIONS:
Drug: Methylprednisolone 40 mg + Ropivacaine + Saline — To infiltrate the study solution, the surgeon will inject the incision site with a 10 cm long, 22-gauge needle before the closing of the incision site. A standard volume of 10 ml in each level will be injected, based on the study by Milligan et al., with a total of 5ml study solution injected laterally into the erector spinae muscle and 5 ml subcutaneously along both margins of the incision. This standardization will be on the basis of the number of levels to be treated, and will be consistent in each patient. The depth of penetration will include the subcutaneous tissues, paravertebral muscles, along with the deep muscles surrounding the spinous process, lamina, transverse process and facet joints; the epidural space and intrathecal space will be spared. The local infiltration solution in the treatment group will consist of a total of 30 ml study solution, containing 1 ml of 40 mg methylprednisolone plus 15ml of 1% ropivacaine and 14 ml saline.
  Arms: methylprednisolone + ropivacaine + saline
Drug: Ropivacaine + Saline — To infiltrate the study solution, the surgeon will inject the incision site with a 10 cm long, 22-gauge needle before the closing of the incision site. A standard volume of 10 ml in each level will be injected, based on the study by Milligan et al., with a total of 5ml study solution injected laterally into the erector spinae muscle and 5 ml subcutaneously along both margins of the incision. This standardization will be on the basis of the number of levels to be treated, and will be consistent in each patient. The depth of penetration will include the subcutaneous tissues, paravertebral muscles, along with the deep muscles surrounding the spinous process, lamina, transverse process and facet joints; the epidural space and intrathecal space will be spared. The local infiltration solution in the control group will consist of a total of 30 ml study solution, containing 15 ml of 1% ropivacaine and 15ml saline.
  Arms: ropivacaine + saline

SUMMARY:
Laminoplasty and laminectomy are useful surgical procedures for the management of various conditions pertaining the spinal cord such as myelopathy, radiculopathy, neoplasm, stenosis, disc herniation, hematoma, abscess, traumatic injuries, etc. Both are generally effective procedures that decompress the spinal cord by expanding the space available for the spinal cord. Both procedures provide good neural decompression and functional improvement after surgery, thereby preventing catastrophic cord injury. However, patients undergoing these procedures experience severe pain in the postoperative period; this may lead to the increase in postoperative morbidity and complications. Suboptimal analgesic therapy causes discomfort to the patient and could increase the incidence of postoperative complications, prolong hospital stay and increase health expenses. The extensive exposure to multiple levels in spine surgeries lead to postoperative pain caused by muscular dissection and requires adequate pain relief to hasten rehabilitation, so that the incidence of chronic pain is significantly decreased. This pain is usually treated with intramuscular, epidural or IV-PCA (Intravenous- Patient Controlled Analgesia) opioids. Several oral analgesics, intermittent intravenous and intramuscular injections and PCA with several systemic side effects, have long been used for the control of postoperative pain. In 1953, Lewis et al. established that local infiltration is a reliable pain relief technique for postoperative pain, with the advantages of safety, simplicity and low cost. The intraoperative injection of 40 mg of methylprednisolone via the intra-buccal approach into the masseter muscle has found to have significantly reduced swelling, trismus and postoperative pain associated with the surgical extraction of impacted lower third molars. A single, preoperative dose of Methylprednisolone 125 mg IV before Total Knee Arthroplasty led to improvement of postoperative analgesia and immediate recovery, when combined with an extensive, multimodal oral and local infiltration analgesic regime. Preemptive administration of bupivacaine or bupivacaine plus methylprednisolone to the paravertebral muscles in patients undergoing lumbar discectomy has been proved to provide effective analgesia in the early postoperative period, when compared to patients who received no local anesthetic or steroid. The infiltration of levobupivacaine and bupivacaine plus methylprednisolone in single distance-single site, lumbar disc surgery established that postoperative analgesic requirement was significantly lower and the first analgesia demand time was also significantly later in the local anesthesia plus methylprednisolone group, compared to the control group. A randomized controlled trial of a larger scale, with a longer follow-up period, could provide a more significant data. Therefore this study has been designed as a prospective, randomized, open-label, blinded endpoint (PROBE) study with a 1 month follow-up period, to compare the efficacy of methylprednisolone plus ropivacaine versus ropivacaine alone, administered before wound closure, for providing analgesia after laminoplasty and laminectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for laminoplasty or laminectomy under general anesthesia
* American Society of Anesthesiologists (ASA) classification I or II
* Age 18 to 64 years

Exclusion Criteria:

* Patient refusal
* Inability to give written informed consent
* Participants who cannot use a patient-controlled analgesia (PCA) device and cannot understand the instructions of a Visual Analogue Score (VAS)
* Previous history of spinal surgery
* Allergy to opioids, methylprednisolone or ropivacaine
* Peri-incisional infection
* History of stroke or a major neurological deficit
* Trauma, deformity
* Psychological problems
* Extreme body mass index (BMI) (< 15 or > 35)
* History of excessive alcohol or drug abuse, chronic opioid use (more than 2 weeks), or use of drugs with confirmed or suspected sedative or analgesic effects
* Patients using systemic steroids
* Pregnant or breastfeeding;
* Preoperative Glasgow Coma Scale < 15
* Participants who have received radiation therapy or chemotherapy preoperatively, or a high probability to require a postoperative radiation therapy or chemotherapy according to the preoperative imaging

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the cumulative sufentanil dose during the 48 hours after surgery via the PCA device. | Within 48 hours after the surgery
  All participates will receive an electronic intravenous patient-controlled analgesia (PCA) device. Participates will be advised to push the analgesic demand button if they feel pain.

SECONDARY OUTCOMES:
Visual Analogue Score | 2 hours, 4 hours, 8 hours, 24 hours, 48 hours, 72 hours, 1 week, 2 weeks and 4 weeks after surgery
  Pain will be assessed by the visual analogue scale (VAS): VAS at movement and VAS at rest in which scores (0 indicates no pain, 10 indicates the most severe pain imaginable, a higher score means worse pain)
Cumulative sufentanil dose for four separate periods | 0-4, 4-8, 8-24, and 24-48 hours
  The cumulative sufentanil dose for four separate periods (0-4, 4-8, 8-24, and 24-48 hours), a total press count including both valid and invalid presses. ( a higher cumulative sufentanil dose means worse pain)
First analgesia demand on the PCA device | Within 48 hours postoperatively
  The time from the end of the surgery to the first administration of analgesia via the PCA device ( a faster analgesia demand means worse pain)
Patient Satisfaction Score | At 2 hours, 4 hours, 8 hours, 24 hours, 48 hours, 72 hours, 1 week, 2 weeks and 4 weeks postoperatively
  Patient Satisfaction Score (PSS) used in this study comprises of points 1-4: 1- Surgery met my expectations; 2- I did not improve as much as I had hoped but I would undergo the same operation for the same results; 3- Surgery helped but I would not undergo the same operation for the same outcome; 4- I am the same or worse as compared to before surgery; ( a higher score means worse pain)
Postoperative Nausea and Vomiting | 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
  Postoperative Nausea and Vomiting (PONV) will be measured using an ordinal scale, with 0 - no nausea; 1 - mild nausea not requiring treatment; 2 - nausea requiring treatment; 3 - vomiting ( a higher score means worse outcome)
Ramsay Sedation Scale | 2 hours, 4 hours, 8 hours, 24 hours, 48 hours after surgery
  Ramsay Sedation Scale (RSS) will be measured using a 6-point scale to assess sedation levels, with 1 indicating agitated, anxious; 2 - cooperative; 3 - only responds to commands; 4 - strong response to glabellar tapping or noisy stimulants; 5 - weak response to glabellar tapping or noisy stimulants; 6 - no response ( a higher score means worse outcome)
The World Health Organization Quality of Life-BREF scores | 4 weeks after surgery
  The World Health Organization Quality of Life-BREF (WHOQOL-BREF) scores will be used to obtain scores for four domains related to quality of life: physical health (7 items), psychological (6 items), social relationships (3 items) and environment (8 items). It will also include two stand-alone questions on overall quality of life and satisfaction with health. Each question will be rated on a scale of 1-5 with higher scores signifying better quality of life.
Oswestry Disability Index | Preoperatively and at 4 weeks postoperatively
  Functional disability will be assessed preoperatively and at 4 weeks after surgery using the Oswestry Disability Index (ODI). It will include 10 questions about pain and activities of daily living. Each item will have five response categories from no pain related disability (0), to the worst possible pain related disability (100) ( a higher score means worse pain)
Patient Scar Assessment and the Observer Scar Assessment Scale | 4 weeks postoperatively
  Patient Scar Assessment and Observer Scar Assessment Scale (POSAS), comprised of subjective symptoms of pain and pruritus, such as vascularity, pigmentation, thickness, relief, pliability, surface area and overall opinion will be assessed at 1 month postoperatively; 0 represents normal skin and 10 represents worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Yoon ST, Hashimoto RE, Raich A, Shaffrey CI, Rhee JM, Riew KD. Outcomes after laminoplasty compared with laminectomy and fusion in patients with cervical myelopathy: a systematic review. Spine (Phila Pa 1976). 2013 Oct 15;38(22 Suppl 1):S183-94. doi: 10.1097/BRS.0b013e3182a7eb7c. PMID 23963000
- [Background] Hardman J, Graf O, Kouloumberis PE, Gao WH, Chan M, Roitberg BZ. Clinical and functional outcomes of laminoplasty and laminectomy. Neurol Res. 2010 May;32(4):416-20. doi: 10.1179/174313209X459084. Epub 2009 Jul 8. PMID 19589202
- [Background] Joshi GP, McCarroll SM, O'Rourke K. Postoperative analgesia after lumbar laminectomy: epidural fentanyl infusion versus patient-controlled intravenous morphine. Anesth Analg. 1995 Mar;80(3):511-4. doi: 10.1097/00000539-199503000-00013. PMID 7864416
- [Background] Kundra P, Gurnani A, Bhattacharya A. Preemptive epidural morphine for postoperative pain relief after lumbar laminectomy. Anesth Analg. 1997 Jul;85(1):135-8. doi: 10.1097/00000539-199707000-00024. PMID 9212136
- [Background] Mesfin A, Park MS, Piyaskulkaew C, Chuntarapas T, Song KS, Kim HJ, Riew KD. Neck Pain following Laminoplasty. Global Spine J. 2015 Feb;5(1):17-22. doi: 10.1055/s-0034-1394297. Epub 2014 Oct 25. PMID 25650126
- [Background] Leslie K, Troedel S, Irwin K, Pearce F, Ugoni A, Gillies R, Pemberton E, Dharmage S. Quality of recovery from anesthesia in neurosurgical patients. Anesthesiology. 2003 Nov;99(5):1158-65. doi: 10.1097/00000542-200311000-00024. PMID 14576554
- [Background] Cherian MN, Mathews MP, Chandy MJ. Local wound infiltration with bupivacaine in lumbar laminectomy. Surg Neurol. 1997 Feb;47(2):120-2; discussion 122-3. doi: 10.1016/s0090-3019(96)00255-8. PMID 9040811
- [Background] LEWIS DL, THOMPSON WA. Reduction of post-operative pain. Br Med J. 1953 May 2;1(4817):973-4. doi: 10.1136/bmj.1.4817.973. No abstract available. PMID 13032582
- [Background] Gurbet A, Bekar A, Bilgin H, Ozdemir N, Kuytu T. Preemptive wound infiltration in lumbar laminectomy for postoperative pain: comparison of bupivacaine and levobupivacaine. Turk Neurosurg. 2014;24(1):48-53. doi: 10.5137/1019-5149.JTN.8431-13.0. PMID 24535791
- [Background] Gurbet A, Bekar A, Bilgin H, Korfali G, Yilmazlar S, Tercan M. Pre-emptive infiltration of levobupivacaine is superior to at-closure administration in lumbar laminectomy patients. Eur Spine J. 2008 Sep;17(9):1237-41. doi: 10.1007/s00586-008-0676-z. Epub 2008 Apr 19. PMID 18425538
- [Background] Esen E, Tasar F, Akhan O. Determination of the anti-inflammatory effects of methylprednisolone on the sequelae of third molar surgery. J Oral Maxillofac Surg. 1999 Oct;57(10):1201-6; discussion 1206-8. doi: 10.1016/s0278-2391(99)90486-x. PMID 10513866
- [Background] Vegas-Bustamante E, Mico-Llorens J, Gargallo-Albiol J, Satorres-Nieto M, Berini-Aytes L, Gay-Escoda C. Efficacy of methylprednisolone injected into the masseter muscle following the surgical extraction of impacted lower third molars. Int J Oral Maxillofac Surg. 2008 Mar;37(3):260-3. doi: 10.1016/j.ijom.2007.07.018. Epub 2008 Mar 4. PMID 18296027
- [Background] Lunn TH, Kristensen BB, Andersen LO, Husted H, Otte KS, Gaarn-Larsen L, Kehlet H. Effect of high-dose preoperative methylprednisolone on pain and recovery after total knee arthroplasty: a randomized, placebo-controlled trial. Br J Anaesth. 2011 Feb;106(2):230-8. doi: 10.1093/bja/aeq333. Epub 2010 Dec 3. PMID 21131371
- [Background] Ersayli DT, Gurbet A, Bekar A, Uckunkaya N, Bilgin H. Effects of perioperatively administered bupivacaine and bupivacaine-methylprednisolone on pain after lumbar discectomy. Spine (Phila Pa 1976). 2006 Sep 1;31(19):2221-6. doi: 10.1097/01.brs.0000232801.19965.a0. PMID 16946657
- [Background] Milligan KR, Macafee AL, Fogarty DJ, Wallace RG, Ramsey P. Intraoperative bupivacaine diminishes pain after lumbar discectomy. A randomised double-blind study. J Bone Joint Surg Br. 1993 Sep;75(5):769-71. doi: 10.1302/0301-620X.75B5.8376436.
- [Background] Mobbs RJ, Li J, Sivabalan P, Raley D, Rao PJ. Outcomes after decompressive laminectomy for lumbar spinal stenosis: comparison between minimally invasive unilateral laminectomy for bilateral decompression and open laminectomy: clinical article. J Neurosurg Spine. 2014 Aug;21(2):179-86. doi: 10.3171/2014.4.SPINE13420. Epub 2014 May 30. PMID 24878273